#### **CONSENT FOR RESEARCH**

Penn State College of Medicine The Milton S. Hershey Medical Center

Title of Project: The Efficacy of Local Anesthetics to Reduce Shoulder Pain Post-Steroid Injections

Principal Investigator: Dr. Robert Gallo

Address: Penn State Milton S. Hershey Medical Center, Bone & Joint Institute, 30 Hope Drive, EC089, PO Box

859, Hershey, PA 17033

Telephone Numbers: Weekdays: 8:00 a.m. to 5:00 p.m. (717) 531-5638.

After hours call (717) 531-8521. Ask for the orthopaedic doctor on 24-hour call.

| Sub | ect's Printed Name: |
|-----|---------------------|

We are asking you to be in a research study.

Whether or not you take part is up to you. You can choose not to take part. You can agree to take part and later change your mind. Your decision will not be held against you.

This form gives you information about the research. Please ask questions about anything that is unclear to you and take your time to make your choice.

#### 1. Why is this research study being done?

We are asking you to be in this research study because your doctor has determined that a steroid injection for the treatment for your shoulder pain is an appropriate intervention.

This research is being done to compare pain relief and efficacy of shoulder injections using one of the following:

- Group A=Injection of 1 ml of 40 mg Kenalog combined with 4 ml of 1% lidocaine
- Group B=Injection of 1 ml of 40 mg Kenalog combined with 4 ml of 1% lidocaine after 2 ml in subcutaneous injection
- Group C=Injection of 1 ml of 40 mg Kenalog combined with 4 ml of 1% lidocaine after applying ethyl chloride spray for 3 seconds

All steroid injections will contain lidocaine in the solution.

The specific aim of this prospective study is to determine whether local anesthetics prior to steroid injections reduce pain and consequently if they are cost-effective in the treatment for shoulder problems.

Approximately 150 people will take part in this research study at Hershey Medical Center.

# 2. What will happen in this research study?

After you have read through this consent form, all of your questions have been answered to your satisfaction, and you have agreed to participate by signing this form, it will be determined by reviewing your medical history if you meet all of the criteria to participate in the study.

If you are eligible to be in the study, you will be randomized (assigned at random, like flipping a coin) to one of three study groups:

- o Group A=Injection of 1 ml of 40 mg Kenalog combined with 4 ml of 1% lidocaine
- Group B=Injection of 1 ml of 40 mg Kenalog combined with 4 ml of 1% lidocaine after 2 ml in subcutaneous injection
- Group C=Injection of 1 ml of 40 mg Kenalog combined with 4 ml of 1% lidocaine after applying ethyl chloride spray for 3 seconds

All steroid injections will contain lidocaine in the solution.

All treatment drugs are FDA approved and considered standard of care.

Randomization means that neither you nor your study doctor will choose what group you will be in. You will have an equal (1 out of 3) chance of being placed in any one of the three groups. The research coordinator will ask you to rate your current pain on a visual pain scale before the injection. Then, the study investigator will perform the injection of your shoulder. Immediately after the injection is finished and ten minutes after the injection, you will be asked to rate your current pain using the same visual pain scale.

#### What are my responsibilities if I take part in this research?

If you take part in this research, your major responsibilities will include:

- Completing the visual pain scale during the visit.
- Allowing access to your medical records as it pertains to this study.

### 3. What are the risks and possible discomforts from being in this research study?

There is a risk of loss of confidentiality if your medical information or your identity are obtained by someone other than the investigators, but precautions will be taken to prevent this from happening. The confidentiality of your electronic data created by you or by the researchers will be maintained to the degree permitted by the technology used. Absolute confidentiality cannot be guaranteed.

You will be assigned to a treatment program by chance. The treatment you receive may prove to be less effective or to have more side effects than the other research treatment(s) or other available treatments.

Ethyl Chloride - freezing may alter skin pigment.

Kenalog - joint tissue damage, swelling in your veins, allergic reaction, infection, increase in blood sugar.

Lidocaine - itching, rash, swelling of the skin, pain at the injection site, numbness, dizziness, and allergic reactions. Rarely, when injected into the blood stream lidocaine can cause confusion, coma, seizures, respiratory arrest, heart beat irregularities, and toxicities; however, in this study lidocaine will not be injected into your bloodstream.

There is risk of some pain and discomfort with the injection as well as the possibility of nerve damage after the injection.

# 4. What are the possible benefits from being in this research study?

## 4a. What are the possible benefits to me?

You may or may not benefit from this particular research study. The treatment group that you are assigned to could be more beneficial than another in providing you pain relief.

## 4b. What are the possible benefits to others?

The results of this study may guide future treatment decisions.

# 5. What other options are available instead of being in this research study?

You do not have to take part in this study to be treated for your condition. Instead of participating in this research, you could:

- Receive commercially available treatments such as a topical anesthetic .
- Be part of a different research study, if one is available.
- Choose not to be treated for your medical condition.

Before you decide if you want to be in this research, we will discuss the other choices that are available to you. We will tell you about the possible benefits and risks of these choices.

The therapy offered in this research is available to you without taking part in this research study.

#### 6. How long will I take part in this research study?

If you agree to take part, it will take you about 10 extra minutes to fill out the questionnaires for the study. Your participation ends with this clinic visit.

## 7. How will you protect my privacy and confidentiality if I decide to take part in this research study?

#### 7a. What happens to the information collected for the research?

Efforts will be made to limit the use and sharing of your personal research information. In our research files at The Milton S. Hershey Medical Center (HMC) and Penn State College of Medicine (PSU) we will include these identifiers: dates, your name, medical record number, phone number, and a code number.

- A list that matches your name with your code number will be kept in a locked file in Dr. Gallo's research office.
- Your research records will be labeled with your code number and kept in a safe area in Dr. Gallo's research office.
- A copy of this signed consent form will be included in your HMC medical record. This means that other HMC healthcare providers will know you are in this study.

In the event of any publication or presentation resulting from the research, no personally identifiable information will be shared.

### 7b. How will my identifiable health information be used?

If you give your consent, health information that can be traced to you will be collected for this research study. In general, under federal law, health information is private. However, there are exceptions to this rule, and you should know who may be able to see, use, and share your health information for research and why they may need to do so.

The research team may use the following health information:

- Past, present, and future medical records
- New health information from tests, procedures, visits, interviews, or forms filled out as part of this research study.

The following people/groups may see, use, and share your identifiable health information:

- HMC/PSU research staff involved in this study
- The HMC/PSU Institutional Review Board (IRB), a group of people who review the research study to protect subjects' rights and welfare
- The HMC/PSU Human Subjects Protection Office
- The HMC/PSU Research Quality Assurance Office
- Non-research staff within HMC/PSU who need this information to do their jobs (such as for treatment, payment (billing), or health care operations)
- Federal and state agencies (such as the U.S. Food and Drug Administration, the Office for Human Research Protections, the Department of Health and Human Services, the National Institutes of Health, and other U.S. or foreign government bodies that oversee or review research)
- The HMC/PSU pharmacy
- Organizations that provide independent accreditation and oversight of hospitals and research
- Public health and safety authorities (for example, if we learn information that could mean harm to you or others, we may need to report this, as required by law)

These groups may also review and/or copy your original PSU/HMC records while looking at the results of the research study. It is possible that some of the other people/groups who receive your health information may not be required by Federal privacy laws to protect your information. We share your information only when we must, and we ask anyone who receives it from us to protect your privacy.

Because research is an ongoing process, your permission for the use, storage and sharing of your health information will continue indefinitely.

#### Your privacy rights:

- You have the right to refuse to sign this form that allows us to use and share your health information for research; however, if you don't sign it, you will not be able to take part in this research study.
- You have the right to withdraw your permission for us to use or share your health information for this research study. If you want to withdraw your permission, you must notify the person in charge of this research study in writing using the address on the front of this form. Once permission is withdrawn, you cannot continue to take part in the study.
- If you withdraw your permission, we will stop collecting health information about you for this study; we may continue to use and share your health information that we already have if it is necessary

for safety and scientific soundness of the research study; and we will not be able to take back information that has already been used or shared with others.

• You have the right to see and get a copy of your health information that is used or shared for treatment or for payment. However, you may not be allowed to see or copy certain health information that is a part of this research study. This is only for the period of the study. You will be allowed to see that information when the entire research study is complete.

## 8. What are the costs of taking part in this research study?

## 8a. What will I have to pay for if I take part in this research study?

For costs of tests and procedures that are only being done for the research study:

- You and/or your insurance company will not be charged for the cost of any tests or procedures that
  are required as part of the research and are outside the standard of care (what is normally done)
  for your condition.
- The research-related tests and procedures that will be provided at no cost to you include: completion of the visual pain scale before and after the standard of care injection.

For costs of medical services for care you would receive even if you were not in this research study:

- You and/or your insurance company will be responsible for the cost of routine medications, tests and procedures that you would receive even if you were not in this research.
- You and/or your insurance company will be billed for the costs of these routine tests and procedures in the usual manner.
- You will be responsible for any co-payments, co-insurance and deductibles that are standard for your insurance coverage.
- You will be responsible for any charges not reimbursed by your insurance company.
- Some insurance companies will not pay for routine costs for people taking part in research studies. Before deciding to be in this research you should check with your insurance company to find out what they will pay for.

If you have any questions about costs and insurance, ask the research study doctor or a member of the research team.

# 8b. What happens if I am injured as a result of taking part in this research study?

It is possible that you could develop complications or injuries as a result of being in this research study. If you experience a side effect or injury and emergency medical treatment is required, seek treatment immediately at any medical facility. If you experience a side effect or injury and you believe that emergency treatment is not necessary, you should contact the principal investigator listed on the first page of this consent form as soon as possible and he/she will arrange for medical treatment.

HMC/PSU compensation for injury

- There are no plans for HMC/PSU to provide financial compensation or free medical treatment for research-related injury.
- If an injury occurs, medical treatment is available at the usual charge.
- Costs will be charged to your insurance carrier or to you.
- Some insurance companies may not cover costs associated with research injuries.
- If these costs are not covered by your insurance, they will be your responsibility.

When you sign this form you are not giving up any legal right to seek compensation for injury.

## 9. Will I be paid to take part in this research study?

You will not receive any payment or compensation for being in this research study.

### 10. Who is paying for this research study?

The institution and investigators are not receiving any funds to support this research study.

## 11. What are my rights if I take part in this research study?

Taking part in this research study is voluntary.

- You do not have to be in this research.
- If you choose to be in this research, you have the right to stop at any time.
- If you decide not to be in this research or if you decide to stop at a later date, there will be no penalty or loss of benefits to which you are entitled.

If you stop being in the research, already collected data may not be removed from the study database. You will be asked whether the investigator can collect medical information from your routine medical care. If you agree, this data will be handled the same as research data. If you withdraw completely from the research study, no further information will be collected and your participation will end. You may discontinue taking part at any time without penalty or loss of benefits to which you are otherwise entitled.

Your research doctor may take you out of the research study without your permission.

- Some possible reasons for this are: continuing the research would be harmful, your condition has become worse, you did not follow the instructions of the study doctor, you experience serious side effects
- If your participation ends early, you may be asked to visit the research doctor for a final visit.

If you will be in another clinical research study at Hershey Medical Center or elsewhere while in this research, you should discuss the procedures and/or treatments with your physician or the study doctors. This precaution is to protect you from possible side effects from interactions of research drugs, treatments or testing.

During the course of the research you will be provided with any new information that may affect your health, welfare or your decision to continue participating in this research.

### 12. If I have questions or concerns about this research study, whom should I call?

Please call the head of the research study, Dr. Robert Gallo at 717-531-5638 or the orthopedic surgery doctor on 24-hour call at 531-8521 if you:

- Have questions, complaints or concerns about the research.
- Believe you may have been harmed by being in the research study.

You may also contact the research protection advocate in the HMC Human Subjects Protection Office (HSPO) at 717-531-5687 if you:

- Have questions regarding your rights as a person in a research study.
- Have concerns or general questions about the research.
- Have questions about your privacy and the use of your personal health information.

• You may also call this number if you cannot reach the research team or wish to talk to someone else about any concerns related to the research.

You may visit the HSPO's web site at http://pennstatehershey.org/irb under subject information for:

Information about your rights when you are in a research study;

Your signature below means that you have explained the research to the subject or subject

- Information about the Institutional Review Board (IRB), a group of people who review the research to protect your rights; and
- Links to the federal regulations and information about the protection of people who are in research studies. If you do not have access to the internet, copies of these federal regulations are available by calling the HSPO at (717) 531-5687.

A description of this clinical trial will be available on http://www.ClinicalTrials.gov, as required by U.S. Law. This Web site will not include information that can identify you. At most, the Web site will include a summary of the results. You can search this Web site at any time.

## INFORMED CONSENT AND AUTHORIZATION TO TAKE PART IN RESEARCH

#### **Signature of Person Obtaining Informed Consent**

| representative and have answer | ed any question | ns he/she h | as about the re | search. |
|---|---|---|---|---|
| Signature of person who explaine (Only approved investigators for | | | Time<br>ne research and | Printed Name obtain informed consent.) |
| Signature of Person Giving Information Discussed this research is Read the information in the Had the opportunity to a Your signature below means the currently have about the research signed and dated form to keep for | t being in this re<br>tudy with an inv<br>this form, and<br>sk any question<br>nat you have r<br>h and those que | esearch you<br>vestigator,<br>s you may h<br>eceived thi<br>estions have | should have: ave. s information, | |
| Signature of Subject | | | | |
| By signing this consent form, you allow your information to be used | • | | • | in this research and agree to |
| Signature of Subject | – ————<br>Date | <u>-</u><br>Ti | <br>me P | Printed Name |